CLINICAL TRIAL: NCT05132868
Title: Assessments of Genetic Counseling Augmented With an Educational Video or Pamphlet Versus Traditional Counseling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, James Ford, Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-61374; VAR0214 (Other: OnCore); NCI-2022-00606 (Other: CTRP)
Record Dates: First submitted 2021-10-25; First posted 2021-11-24 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Quality; Prostate Cancer; Gastrointestinal Cancer; Gynecologic Cancer; Ovarian Cancer; Pancreatic Cancer
Keywords: cancer genetic counseling; educational video; pamphlet
MeSH Terms: conditions — Prostatic Neoplasms; Gastrointestinal Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pre-educated with educational video (Experimental): Participants will receive a message to view educational videos prior to their genetic counseling appointment if they are assigned to a pre-educated arm. The video will be shared with patients via MyHealth in the "education" tab in advance of the genetic counseling session
  Interventions: Other: Educational video and pamphlet; Other: Traditional genetic counseling
- pre-educated with pamphlet (Experimental): Participants will receive a message to view a pamphlet prior to their genetic counseling appointment if they are assigned to a pre-educated arm. The pamphlet will be sent to patients who cannot access the video via regular mail in advance of the genetic counseling session
  Interventions: Other: Educational video and pamphlet; Other: Traditional genetic counseling
- educated during the session (Other): Participants will receive traditional genetic counseling. . After the genetic counseling session, they will fill out a validated survey called the Multi-dimensional Measure of Informed Choice (MMIC) that assesses attitudes, knowledge, and uptake of genetic testing
  Interventions: Other: Traditional genetic counseling

INTERVENTIONS:
Other: Educational video and pamphlet — The primary intervention in this study is watching the video or reading the pamphlet in advance of the genetic counseling session, which overview the same information that we currently provide in-person/via telehealth during the genetic counseling session.
  Arms: pre-educated with educational video; pre-educated with pamphlet
Other: Traditional genetic counseling — Patients will receive traditional genetic counseling

SUMMARY:
The purpose of this research study is to understand the impact of an educational video or pamphlet on the patient experience in a hereditary cancer genetic counseling program. In order to make this assessment, it is necessary to perform qualitative and quantitative research among patients in a hereditary cancer genetic counseling clinic.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for: Limited English Proficiency (LEP), primarily Spanish speaking cohort

* Preferred language for receiving medical information is Spanish
* Has a personal or family history of cancer
* If assigned to the arm where they need to be pre-educated with a video or pamphlet, attests that they viewed the video or pamphlet

Inclusion criteria for: Individuals with a personal or family history of breast cancer cohort

* Personal or family history of breast cancer
* English is preferred language
* If assigned to the arm where they need to be pre-educated with a video or pamphlet, attests that they viewed the video or pamphlet

Inclusion criteria for: Individuals with a personal or family history of prostate cancer cohort

* Personal or family history of prostate cancer
* English is preferred language
* If assigned to the arm where they need to be pre-educated with a video or pamphlet, attests that they viewed the video or pamphlet

Inclusion criteria for: Individuals with a personal or family history of any type of cancer referred for germline testing based on a genetic variant identified during tumor genomic analysis for the patient or affected family member cohort.

* Personal or family history of any type of cancer
* Referred based on a variant identified during tumor genomic analysis
* English is preferred language
* If assigned to the arm where they need to be pre-educated with a video or pamphlet, attests that they viewed the video or pamphlet

Inclusion criteria for: Individuals with a personal or family history of gastrointestinal or gynecologic cancer, referred because they or their affected relative screened positive for Lynch Syndrome based on either an immunohistochemistry test or evidence of mismatch repair deficiency in their tumor cohort.

* Personal or family history of gastrointestinal or gynecologic cancer
* Screened positive for Lynch Syndrome based on IHC or MMR testing
* English is preferred language
* If assigned to the arm where they need to be pre-educated with a video or pamphlet, attests that they viewed the video or pamphlet

Inclusion criteria for: Individuals with a personal or family history of ovarian and/or pancreatic cancer cohort

* Personal or family history of ovarian, and/or pancreatic cancer
* English is preferred language
* If assigned to the arm where they need to be pre-educated with a video or pamphlet, attests that they viewed the video or pamphlet

Exclusion Criteria:

* Individuals who are minors
* Individuals who are decisionally impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Patient impact with educational information prior to genetic counseling | 36 months
  Impact will be defined as the number of questions asked by patient during the counseling.
Patient impact without any educational information prior to genetic counseling | 36 months
  Impact will be defined as the number of questions asked by patient during the counseling.

CONTACTS AND LOCATIONS:
Overall Officials: James Ford, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States